CLINICAL TRIAL: NCT07086560
Title: PERceptions of Diltiazem Versus ADEnosine for Treatment of Supraventricular Tachycardia in the Emergency Department: PERVADE-ED Study
Brief Title: PERceptions of Diltiazem Versus ADEnosine for Treatment of Supraventricular Tachycardia in the Emergency Department
Acronym: PERVADE-ED
Status: Recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Anne E. Zepeski, Clinical Assistant Professor, University of Iowa
Other Study IDs: 202411431
Record Dates: First submitted 2025-04-04; First posted 2025-07-25 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Supraventricular Tachycardia (SVT)
Keywords: diltiazem; adenosine; emergency medicine; supraventricular tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Adenosine; Diltiazem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adenosine
  Interventions: Drug: IV adenosine
- Diltiazem
  Interventions: Drug: IV diltiazem

INTERVENTIONS:
Drug: IV adenosine — Patients will not be randomized to intervention but will be categorized based on the exposure of IV adenosine for treatment of SVT received prior to study enrollment
  Groups: Adenosine
Drug: IV diltiazem — Patients will not be randomized to intervention but will be categorized based on the exposure of IV diltiazem for treatment of SVT received prior to study enrollment
  Groups: Diltiazem

SUMMARY:
Supraventricular tachycardia (SVT) is a dysrhythmia characterized rapid heart rate, typically with rapid onset. SVT accounts for over 50,000 emergency department visits per year. Of patients with regular, narrow-complex SVT, the mainstay of therapy includes adenosine and diltiazem. Adenosine is recommend by American and European guidelines as first-line therapy, however adenosine carries unique side effects that are potentially distressing to patients, including: "feeling of impending death or doom", flushing, anxiety, shortness of breath, and chest discomfort. Diltiazem does not carry this side effect profile, but has typically been reserved as second-line treatment due to side effects of low blood pressure associated with this class of medications. Diltiazem and adenosine have not been well studied head-to-head to compare safety and efficacy of their treatment for SVT. The purpose of this study is to evaluate safety and efficacy of adenosine and diltiazem for SVT in the ED (as completed through chart review of specific patient-level outcomes) and capture patient and clinician perspectives of medication satisfaction (through administration of questionnaires).

ELIGIBILITY:
Inclusion Criteria:

1. ED encounter for acute SVT
2. Age >/= 18 years
3. Receipt of IV adenosine and/or IV diltiazem for SVT in the ED or prehospital setting

Exclusion Criteria:

1. Neurologic status precluding survey participation due to medical instability
2. Pregnant
3. Incarcerated
4. Non-English speaking

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years of age) treated for SVT in the ED. The investigators will screen a convenience sample of adult patients presenting with stable SVT in the ED for study eligibility while study investigators (most often emergency medicine clinical pharmacists) are available to enroll participants and administer study questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with SVT treatment | Primary outcome will be assessed during ED visit
  Patient satisfaction with treatment will be assessed using a Likert scale questionnaire of 1-5. Participants will indicate their satisfaction with treatment by indicating a score of 1-5, 1 being "not at all satisfied" and 5 being "extremely satisfied".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No